CLINICAL TRIAL: NCT01893281
Title: The Effect of Testosterone Topical Solution (LY900011) in Hypogonadal Men With Suboptimal Response to a Topical Testosterone Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14980; I5E-US-TSBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topical Testosterone Solution (Experimental): Topical Testosterone Solution 30 milligrams up to 120 milligrams per day (mg/day) administered topically to axillae titrated based on testosterone levels.
  Interventions: Drug: Topical Testosterone Solution

INTERVENTIONS:
Drug: Topical Testosterone Solution — Administered topically to axillae.
  Other Names: LY900011; Axiron; Testosterone Solution 2%

SUMMARY:
This study will evaluate if testosterone solution can raise testosterone hormone levels into the normal range after treatment for up to 9 Weeks, in those participants with a documented history of subtherapeutic levels [total testosterone <300 nanograms per deciliter (ng/dL)] when previously treated with a topical testosterone gel.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and provide signed informed consent before starting trial activities related to this study (including discontinuing testosterone replacement therapy prior to Screening)
* Male participants with a diagnosis of hypogonadism and documented biochemical failure (total testosterone <300 ng/dL) when treated with the highest dose of a topical testosterone gel tolerated by the participant. Documentation of biochemical failure includes: the name and dose of the topical testosterone gel, a lab report showing a total testosterone level <300 ng/dL while on therapy, or a written chart report stating that there was a clear lack of efficacy, including the participant's serum total testosterone level at the time of failure
* Screening serum total testosterone level of <300 ng/dL (based on the average of 2 morning blood samples taken at least 30 minutes apart) at Screening
* Prostate Specific Antigen (PSA) <4 nanogram per milliliter (ng/mL) at Screening
* If the participant is receiving testosterone replacement therapy and is willing to discontinue testosterone replacement therapy to enter the study, their screening total testosterone level cannot be checked until at least 14 days after discontinuing topical therapies, or after at least 28 days for participants using short-acting intramuscular (IM) therapies

Exclusion Criteria:

* Any previous treatment with testosterone topical solution (LY900011)
* Known or suspected carcinoma (or history of carcinoma) of the prostate or suspicious nodules on digital rectal exam at Screening
* Known or suspected breast cancer or history of breast cancer
* Severe sleep apnea (untreated or unsuccessfully treated) in the opinion of the study investigator
* Use of long-acting IM testosterone undecanoate in the 6-month period prior to Screening
* History of the use of an implanted testosterone pellets (Testopel)
* International Prostate Symptom Score (IPSS) total score >19 at Screening
* Hematocrit ≥50% at Screening. For sites located at elevations ≥4500 feet, participants will be excluded with hematocrit >54% according to investigator discretion. Any participant with a hematocrit >54% at later study visits will be withdrawn from the study
* Significant history of allergy and/or sensitivity to the drug products or excipients, including any history of sensitivity to testosterone and/or sunscreens
* Dermatologic condition in underarm area that might interfere with testosterone absorption (for example, eczema) or that could be exacerbated by topical testosterone replacement therapy
* History of luteinizing hormone-releasing hormone (LHRH) antagonist or agonist treatment in the 6 months prior to Screening
* Exhibit any evidence of congestive heart failure [New York Heart Association (NYHA) Class 2 or above] within 6 months prior to Screening
* Exhibit evidence of severe renal impairment [creatinine clearance <30 milliliter per minute (mL/min) as determined by the Cockcroft-Gault formula] at Screening
* Exhibit a history of severe liver disease or clinical evidence of hepatic impairment at Screening
* Any condition that would interfere with the participant's ability to provide informed consent, or comply with study instructions, or would place the participant at increased risk, or might confound the interpretation of the study results
* Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device (other than the investigational product used in this study), or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (21):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Encinitas, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parker, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coeur d'Alene, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anderson, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeffersonville, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elkhorn, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marlton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden City, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poughkeepsie, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cary, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salisbury, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshall, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Testosterone Solution: Testosterone, initially 60 milligrams (mg) once daily (QD), titrated to effect as needed (range 30-120 mg QD), administered as a 2% topical solution for up to 9 weeks.
Period: Overall Study
Arm/Group | Topical Testosterone Solution
Started | 78
Received at Least 1 Dose of Study Drug | 78
Completed | 75
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Topical Testosterone Solution: Testosterone, initially 60 mg QD, titrated to effect as needed (range 30-120 mg QD), administered as a 2% topical solution for up to 9 weeks.
Arm/Group | Topical Testosterone Solution
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 73
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Normal Serum Testosterone Levels
Description: Normal serum testosterone level is defined as ≥300 to ≤1050 nanograms/deciliter (ng/dL). Serum testosterone levels were measured by liquid chromatography and tandem mass spectrometry (LC/MS-MS). Percentage of participants = (number of participants who achieved normal serum testosterone level) / (number of treated participants who had serum testosterone level measured) * 100.
Time Frame: Baseline through Study Completion (Up to 9 Weeks)
Population: All enrolled participants who received at least 1 dose of study drug and had serum testosterone level measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Topical Testosterone Solution
Number analyzed (Participants) | 76
percentage of participants | 94.7 [87 to 99]

2. Secondary Outcome: Change From Baseline in Serum Testosterone Levels
Description: Serum testosterone levels were measured by LC/MS-MS.
Time Frame: Baseline, Study Completion (Up to 9 Weeks)
Population: All enrolled participants who received at least 1 dose of study drug with non-missing data at baseline and at least 1 post baseline measurement. Last-observation-carried-forward (LOCF) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Topical Testosterone Solution
Number analyzed (Participants) | 76
ng/dL | 354.8 (280.99)
Statistical Analysis 1: Comparison: Topical Testosterone Solution; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Participants in Each Category of the Patient Global Impression - Improvement (PGI-I) Scale for Sexual Drive
Description: PGI-I for sexual drive is a participant-rated questionnaire that measure change in sexual drive after a participant begins the study drug. The questionnaire was completed at every visit post baseline using a 7-point scale where a score of 1 indicated that the participant's sexual drive was "very much better," a score of 4 indicated that the participant had experienced "no change" in sexual drive and a score of 7 indicated that the participant's sexual drive was "very much worse". Percentage of participants = (number of participants in the category) / (total number of participants who responded to the questionnaire) * 100.
Time Frame: Study Days 15, 22, 36, 43, 57, 64 and endpoint
Population: All enrolled participants who received at least 1 dose of study drug and responded to PGI-I sexual drive questionnaire at specified time points. Endpoint is defined as the last non-missing PGI-I scale for sexual drive collected from Day 15 through end of study.
Measure: Number; unit: percentage of participants
Arm/Group | Topical Testosterone Solution
Number analyzed (Participants) | 77
percentage of participants
  Very much better - Day 15 (n=76) | 3.95
  Much better - Day 15 (n=76) | 11.84
  A little better - Day 15 (n=76) | 44.74
  No change - Day 15 (n=76) | 38.16
  A little worse - Day 15 (n=76) | 1.32
  Much worse - Day 15 (n=76) | 0.00
  Very much worse - Day 15 (n=76) | 0.00
  Very much better - Day 22 (n=76) | 5.26
  Much better - Day 22 (n=76) | 25.00
  A little better - Day 22 (n=76) | 39.47
  No change - Day 22 (n=76) | 30.26
  A little worse - Day 22 (n=76) | 0.00
  Much worse - Day 22 (n=76) | 0.00
  Very much worse - Day 22 (n=76) | 0.00
  Very much better - Day 36 (n=22) | 0.00
  Much better - Day 36 (n=22) | 22.73
  A little better - Day 36 (n=22) | 45.45
  No change - Day 36 (n=22) | 31.82
  A little worse - Day 36 (n=22) | 0.00
  Much worse - Day 36 (n=22) | 0.00
  Very much worse - Day 36 (n=22) | 0.00
  Very much better - Day 43 (n=22) | 4.55
  Much better - Day 43 (n=22) | 22.73
  A little better - Day 43 (n=22) | 36.36
  No change - Day 43 (n=22) | 31.82
  A little worse - Day 43 (n=22) | 4.55
  Much worse - Day 43 (n=22) | 0.00
  Very much worse - Day 43 (n=22) | 0.00
  Very much better - Day 57 (n=6) | 0.00
  Much better - Day 57 (n=6) | 50.00
  A little better - Day 57 (n=6) | 0.00
  No change - Day 57 (n=6) | 50.00
  A little worse - Day 57 (n=6) | 0.00
  Much worse - Day 57 (n=6) | 0.00
  Very much worse - Day 57 (n=6) | 0.00
  Very much better - Day 64 (n=6) | 16.67
  Much better - Day 64 (n=6) | 33.33
  A little better - Day 64 (n=6) | 0.00
  No change - Day 64 (n=6) | 50.00
  A little worse - Day 64 (n=6) | 0.00
  Much worse - Day 64 (n=6) | 0.00
  Very much worse - Day 64 (n=6) | 0.00
  Very much better - Endpoint (n=77) | 7.79
  Much better - Endpoint (n=77) | 27.27
  A little better - Endpoint (n=77) | 35.06
  No change - Endpoint (n=77) | 28.57
  A little worse - Endpoint (n=77) | 1.30
  Much worse - Endpoint (n=77) | 0.00
  Very much worse - Endpoint (n=77) | 0.00

4. Secondary Outcome: Percentage of Participants in Each Category of the Patient Global Impression - Improvement (PGI-I) Scale for Energy Level
Description: PGI-I for energy level is a participant-rated questionnaire that measures change in energy level after a participant begins the study drug. The questionnaire was completed at every visit post baseline using a 7-point scale where a score of 1 indicated that the participant's energy level was "very much better," a score of 4 indicated that the participant had experienced "no change" in energy level and a score of 7 indicated that the participant's energy level was "very much worse". Percentage of participants = (number of participants in the category) / (total number of participants who responded to the questionnaires) * 100.
Time Frame: Study Days 15, 22, 36, 43, 57, 64 and endpoint
Population: All enrolled participants who received at least 1 dose of study drug and responded to PGI-I energy level questionnaire at specified time points. Endpoint is defined as the last non-missing PGI-I scale for energy level collected from Day 15 through end of study.
Measure: Number; unit: percentage of participants
Arm/Group | Topical Testosterone Solution
Number analyzed (Participants) | 77
percentage of participants
  Very much better - Day 15 (n=75) | 4.00
  Much better - Day 15 (n=75) | 16.00
  A little better - Day 15 (n=75) | 44.00
  No change - Day 15 (n=75) | 36.00
  A little worse - Day 15 (n=75) | 0.00
  Much worse - Day 15 (n=75) | 0.00
  Very much worse - Day 15 (n=75) | 0.00
  Very much better - Day 22 (n=76) | 7.89
  Much better - Day 22 (n=76) | 27.63
  A little better - Day 22 (n=76) | 40.79
  No change - Day 22 (n=76) | 22.37
  A little worse - Day 22 (n=76) | 1.32
  Much worse - Day 22 (n=76) | 0.00
  Very much worse - Day 22 (n=76) | 0.00
  Very much better - Day 36 (n=22) | 4.55
  Much better - Day 36 (n=22) | 18.18
  A little better - Day 36 (n=22) | 50.00
  No change - Day 36 (n=22) | 22.73
  A little worse - Day 36 (n=22) | 4.55
  Much worse - Day 36 (n=22) | 0.00
  Very much worse - Day 36 (n=22) | 0.00
  Very much better - Day 43 (n=22) | 4.55
  Much better - Day 43 (n=22) | 27.27
  A little better - Day 43 (n=22) | 40.91
  No change - Day 43 (n=22) | 22.73
  A little worse - Day 43 (n=22) | 4.55
  Much worse - Day 43 (n=22) | 0.00
  Very much worse - Day 43 (n=22) | 0.00
  Very much better - Day 57 (n=6) | 0.00
  Much better - Day 57 (n=6) | 33.33
  A little better - Day 57 (n=6) | 50.00
  No change - Day 57 (n=6) | 16.67
  A little worse - Day 57 (n=6) | 0.00
  Much worse - Day 57 (n=6) | 0.00
  Very much worse - Day 57 (n=6) | 0.00
  Very much better - Day 64 (n=6) | 16.67
  Much better - Day 64 (n=6) | 16.67
  A little better - Day 64 (n=6) | 33.33
  No change - Day 64 (n=6) | 33.33
  A little worse - Day 64 (n=6) | 0.00
  Much worse - Day 64 (n=6) | 0.00
  Very much worse - Day 64 (n=6) | 0.00
  Very much better - Endpoint (n=77) | 10.39
  Much better - Endpoint (n=77) | 29.87
  A little better - Endpoint (n=77) | 35.06
  No change - Endpoint (n=77) | 22.08
  A little worse - Endpoint (n=77) | 2.60
  Much worse - Endpoint (n=77) | 0.00
  Very much worse - Endpoint (n=77) | 0.00

ADVERSE EVENTS:
Arm/Group | Topical Testosterone Solution
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 22/78
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Testosterone Solution (N=78)
Nausea (Gastrointestinal disorders) | 1 (1)
Application site pain (General disorders) | 2 (2)
Influenza like illness (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Allergy to animal (Immune system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood pressure diastolic abnormal (Investigations) | 1 (1)
Blood pressure diastolic decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Heart rate increased (Investigations) | 2 (2)
Weight increased (Investigations) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Testicular atrophy (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days